CLINICAL TRIAL: NCT05835479
Title: A Phase 2, Proof-of-Concept, Multicentre, Open-Label, Randomised, Active-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Rezafungin Combined With 7 Days of Co-Trimoxazole Versus Co-Trimoxazole Monotherapy in HIV-Infected Adults With Pneumocystis Jirovecii Pneumonia
Brief Title: Rezafungin for Treatment of Pneumocystis Pneumonia in HIV Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR907-2501
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Pneumocystis Pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Rezafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rezafungin Acetate /Co-trimoxazole (Experimental): Rezafungin: Weekly intravenous infusion with a loading dose of 400 mg over 1 hour (±10 minutes) on Day 1 followed by maintenance doses of 200 mg over 1 hour (±10 minutes) on Day 8 and Day 15.
  From Day 1 to Day 7, co-trimoxazole will also be given with trimethoprim 15-20 mg/kg/day and sulfamethoxazole 75-100 mg/kg/day.
  For participants with a creatinine clearance between 15 mL/min and 30 mL/min, the dose of co-trimoxazole should be reduced to trimethoprim 7.5-10 mg/kg/day and sulfamethoxazole 37.5-50 mg/kg/day
  Interventions: Drug: Rezafungin Acetate / Co Trimoxazole
- Co-trimoxazole (Active Comparator): From Day 1 to Day 21, co-trimoxazole will be given with trimethoprim 15-20 mg/kg/day and sulfamethoxazole 75-100 mg/kg/day.
  For participants with a creatinine clearance between 15 mL/min and 30 mL/min, the dose of co-trimoxazole should be reduced to trimethoprim 7.5-10 mg/kg/day and sulfamethoxazole 37.5-50 mg/kg/day
  Interventions: Drug: Co-Trimoxazole

INTERVENTIONS:
Drug: Co-Trimoxazole — Oral co-trimoxazole or Intravenous (IV) co-trimoxazole for infusion. Anti fungal medication
  Arms: Co-trimoxazole
Drug: Rezafungin Acetate / Co Trimoxazole — Rezafungin for infusion. Intravenous anti fungal therapy
  Oral co-trimoxazole or Intravenous (IV) co-trimoxazole for infusion. Anti fungal medication
  Arms: Rezafungin Acetate /Co-trimoxazole

SUMMARY:
This study aims to generate clinical data on the efficacy, safety, and tolerability of rezafungin combined with 7 days of co-trimoxazole for treatment of Pneumocystis pneumonia (PCP) in adults living with human immunodeficiency virus (HIV), which would expand the knowledge of clinical use of rezafungin.

DETAILED DESCRIPTION:
The study comprises a Screening period from Day -2 to Day -1, a Treatment period from Day 1 to Day 21, and a Follow-up visit on Day 50 (±2 days). The total duration for the study will be up to approximately 52 days.

Participants meeting the eligibility criteria will be randomised in a 1:1 ratio to either the rezafungin/co-trimoxazole group or co-trimoxazole monotherapy group. Randomisation will be stratified by disease severity into two categories (mild or moderate-to-severe).

After completion of the 21-day treatment, co-trimoxazole for secondary prophylaxis against P. jirovecii will be given to all participants. In participants who are discovered to have an allergy or intolerance to co-trimoxazole during the study, an alternative secondary prophylaxis will be provided as per local practice and treatment guidelines, decided by the treating physician. Participants will have a Follow-up visit on Day 50 (±2 days) to evaluate AEs, treatment response, and rates of PCP relapse or paradoxical IRIS (Immune reconstitution inflammatory syndrome).

Participants will be monitored for AEs from the time the first dose of the study drugs is administered to the Follow-up visit on Day 50 (±2 days). Additional safety assessments including vital signs, safety laboratory evaluations (haematology, serum chemistry panel, and urinalysis), physical examinations (complete and symptom-directed), and 12-lead ECGs will also be assessed. Prior and concomitant medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age.
2. Tested positive for HIV by either blood antigen/antibody combination HIV-1/2 immunoassay, HIV-1/HIV-2 antibody differentiation immunoassay, or nucleic acid tests (e.g., HIV ribonucleic acid [RNA] polymerase chain reaction [PCR]). Participants who are newly diagnosed with HIV infection by an antigen/antibody combination HIV-1/2 immunoassay are allowed to be included in the study, but the infection should be subsequently confirmed by an HIV-1/HIV-2 antibody differentiation immunoassay or nucleic acid tests.
3. Diagnosed with definitive, presumptive, or clinically suspected PCP prior to randomisation.
4. Willing and able to provide written informed consent. If the participant is unable to provide consent, a legally acceptable representative (i.e., acceptable to ICH and local law, as applicable) must provide informed consent on the participant's behalf.
5. Participants of childbearing potential (all biologically female participants between 18 years and <2 years post-menopausal unless surgically sterile) must agree to use a highly effective contraceptive measure during the study period (from enrolment) and for at least 30 days after the last dose of rezafungin.
6. Biologically male participants who are not vasectomised must agree to the following requirements during the study period (from enrolment) and for at least 120 days after the last dose of rezafungin:

   * Refrain from donating sperm PLUS, either
   * Abstain from sexual intercourse with a female of childbearing potential as their preferred and usual lifestyle OR
   * Use barrier contraception (i.e., male condom with or without spermicide) when having sexual intercourse with a female of childbearing potential who is not currently pregnant.

Exclusion Criteria:

1. Under 18 years of age.
2. Known or suspected hypersensitivity or allergic reaction to co-trimoxazole, rezafungin, any echinocandin, or any component of these formulations, including, but not limited to, anaphylaxis or exfoliative skin disorders (e.g., Stevens-Johnson syndrome or toxic epidermal necrolysis).
3. Any contraindication to co-trimoxazole or intake of a medication or supplement known to severely interact with co-trimoxazole as detailed in the Summary of Product Characteristics (SmPC) of co-trimoxazole, including, but not limited to, acute porphyria or a history of drug-induced immune thrombocytopaenia with use of trimethoprim and/or sulphonamides.
4. Creatinine clearance <15 mL/min or receiving renal replacement therapy.
5. Severe hepatic impairment, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 × upper limits of normal (ULN), or total bilirubin >3 × ULN, or a history of chronic cirrhosis (Child-Pugh score >9).
6. A neutrophil count <1,000 cells/µL or a platelet count <50,000 cells/µL.
7. Immunosuppressive disease other than HIV / acquired immunodeficiency syndrome (AIDS) (e.g., haematopoietic stem cell transplant, solid organ transplant, or primary immune deficiencies) OR prolonged use of immune-weakening medications:

   * Having received corticosteroids equivalent to prednisone ≥20 mg daily for at least 14 consecutive days within 30 days prior to study entry, or
   * Having received biologics (e.g., infliximab, ustekinumab), immunomodulators (e.g., methotrexate, mercaptopurine, azathioprine), or cancer chemotherapy within 90 days prior to study entry.
8. Previously diagnosed with PCP and having received treatment in the past 6 weeks.
9. Receiving therapy for PCP at approved therapeutic doses for >48 hours before randomisation. Exception: receipt of an anti-PCP drug at prophylactic doses (i.e., lower than approved therapeutic doses).
10. Meeting National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 criteria for ataxia, tremors, motor neuropathy, or sensory neuropathy of Grade 2 or higher.
11. History of severe ataxia, tremors, or neuropathy or a diagnosis of multiple sclerosis or a movement disorder (including Parkinson's disease and Huntington's disease).
12. Planned or ongoing therapy at Screening with a known severe neurotoxic medication or with a known moderate neurotoxic medication in a participant with ataxia, tremors, motor neuropathy, or sensory neuropathy of NCI-CTCAE version 5.0 Grade 1 or higher.
13. Previous participation in this or any other rezafungin study.
14. Female participants who are pregnant or lactating.
15. Having a concomitant disease or any medical condition (including other HIV-associated infection or complication) that, in the opinion of the Investigator, could pose undue risk to the participant, impede completion of the study procedures (e.g., patients who are not expected to survive even with treatment), or would compromise the validity of the study measurements.
16. Receipt of an investigational drug within 30 days prior to dosing of the study drug(s), presence of an investigational device at the time of Screening, or is planning to participate in another interventional clinical study while enrolled in this study.
17. The Investigator is of the opinion the participant should not participate in the study.

Late Exclusion Criteria:

The diagnosis of PCP will be reviewed by the Investigator on Day 8 (before dosing the study drug). Participants will be withdrawn from the study if any of the following criteria apply (i.e., participants without a diagnosis of definitive or presumptive PCP on Day 8):

1. Lack of positive P. jirovecii immunofluorescence or PCR of bronchoalveolar lavage, endotracheal aspirates, bronchoscopic tissue biopsy, or induced sputum AND serum β-D-glucan below the positive cut-off value.
2. Serum β-D-glucan below the positive cut-off value in participants in whom collection of a suitable respiratory sample is not possible.
3. Radiographic features on chest CT performed after randomisation not consistent with PCP after taking into account the clinical and microbiological findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Therapeutic failure on Day 8 | 8 days
  Therapeutic failure on Day 8, defined by one of the following and confirmed by an independent, blinded Data Review Committee (DRC):
  * Clinical deterioration. The deterioration cannot be solely explained by other infections or causes and is defined as an increase in score of 2 points or more from the score prior to randomisation on Day 1 on the Ordinal Scale for Clinical Improvement (OSCI), as assessed by the Investigator.
  * Requirement for alternative primary therapy for PCP, or intensification of corticosteroid therapy, due to lack of efficacy (as assessed by the Investigator).
  * Death from any cause.

SECONDARY OUTCOMES:
Therapeutic failure at any time during the treatment period (from Day 1 to Day 21) | 21 days
  Therapeutic failure at any time during the treatment period (from Day 1 to Day 21) defined by one of the following and confirmed by an independent, blinded Data Review Committee (DRC):
  * Clinical deterioration. The deterioration cannot be solely explained by other infections or causes and is defined as an increase in score of 2 points or more from the score prior to randomisation on Day 1 on the Ordinal Scale for Clinical Improvement (OSCI), as assessed by the Investigator.
  * Requirement for alternative primary therapy for PCP, or intensification of corticosteroid therapy, due to lack of efficacy (as assessed by the Investigator).
  * Death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Joshi, MD, Study Director — Mundipharma Research Limited
Locations (6):
- South Africa (6):
  - University of Cape Town, Cape Town
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Helen Joseph Hospital, Johannesburg
  - Global Clinical Trials - Pretoria, Pretoria
  - Steve Biko Academic Hospital, Pretoria
  - Netcare Umhlanga Medical Centre, Umhlanga

REFERENCES:
- [Derived] Peghin M, Fishman JA, Grossi PA. Pneumocystis jiroveci: still troublesome to diagnose and treat. Curr Opin Infect Dis. 2025 Oct 18. doi: 10.1097/QCO.0000000000001155. Online ahead of print. PMID 41151592